CLINICAL TRIAL: NCT00464100
Title: Neurodevelopmental Outcomes and Postoperative Hemodynamics in Children With Hypoplastic Left Heart Syndrome
Brief Title: Near-infrared Spectroscopy (NIRS) Neurodevelopmental Outcomes
Acronym: NIRS-ND
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Nancy Ghanayem, Associate Professor, Pediatrics, Critical Care, Medical College of Wisconsin
Other Study IDs: CHW 06/36
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Neurodevelopmental outcomes; congenital heart disease; NIRS monitoring; hypoxia
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We believe that how a baby with Hypoplastic Left Heart Syndrome (HLHS)does after a major open heart operation, measured by things like blood pressure, oxygen saturation, heart rate and others, may have an impact on development. Studying how post-operative condition impacts outcomes may help us to protect babies better when they undergo surgery.

This study will look at some of the long-term outcomes of children with HLHS, including both mental development and quality of life. We will use information from your child's medical record to see if early oxygen delivery has an impact on later development.

DETAILED DESCRIPTION:
Over the past twenty years, the field of congenital heart disease has been marked by globally improved survival after complex congenital heart surgery. These improved results are clearly multi-factorial and include advances in diagnostic technologies, surgical techniques, perfusion strategies, pharmacologic therapies and perioperative monitoring of tissue oxygen delivery.

Hypoplastic left heart syndrome (HLHS) represents an extreme form of complex congenital heart disease in which the infant has prolonged cyanosis and a single systemic right ventricle. Staged palliation beginning with surgery in the neonatal period is the most common approach to infants with HLHS. After initial surgical palliation, infants are critically ill due to ischemia/reperfusion injury from cardiopulmonary bypass, coronary ischemia attributed to diastolic runoff, reduced total ventricular mass, continued hypoxemia during a time of increased metabolic demands, and finally, the inherent inefficiency of parallel circulation. The presence of any one of these physiologic derangements places the infant with HLHS at great risk for ischemia, organ dysfunction, circulatory collapse and, even, death. Postoperative monitoring of venous oximetry and, more recently, near infrared spectroscopy, have identified periods of impaired oxygen delivery and ischemia, allowed for interventions that enhance oxygen delivery and improved survival after cardiac surgery. Although, an apparent relationship exists between oxygen delivery and survival after cardiac surgery, little data is available on the relationship between oxygen delivery and neurodevelopmental outcomes (inclusive of neurocognitive and neuropsychologic outcomes).

Preliminary data from our center has recently identified that reduced venous oximetry was associated with adverse neurodevelopmental outcome. These initial findings warrant further investigation of neurologic injury, specifically, how such morbidity relates to perioperative ischemia and cerebral oxygen delivery. Hence, the purpose of this study is to understand the relationship of perioperative tissue dysoxia and long-term neurodevelopmental morbidity in children subject to oxygen delivery at which neurodevelopment is compromised. Identification of a critical threshold that may be devastating to a child's neurodevelopment and quality of life would allow for early intervention, goal-directed therapy and ultimately, improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* clinical diagnosis of hypoplastic left heart syndrome, status post Norwood procedure, bidirectional Glenn, and completion Fontan, ages 4-5 years old, English-speaking patient and parent, informed consent

Controls:

Healthy children 4-5 years old, English-speaking patient and parent, informed consent

Exclusion Criteria:

* Congenital or acquired abnormality associated with neurologic morbidity independent of cardiac lesion

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases:
  * clinical diagnosis of hypoplastic left heart syndrome, status post Norwood procedure, bidirectional Glenn, and completion Fontan, ages 4-5 years old, English-speaking patient and parent, informed consent
  Controls:
  Healthy children 4-5 years old, English-speaking patient and parent, informed consent
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2013-12-04 (Actual); Study Completion 2013-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ghanayem, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States